CLINICAL TRIAL: NCT00581178
Title: Study to Determine if There Are Specific Clinical Factors to Determine Stent Encrustation
Status: Terminated | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Labcorp Corporation of America Holdings, Inc (Industry)
Responsible Party: Principal Investigator, Victor Huynh, Urology Account Contact, University of California, Irvine
Other Study IDs: 2007-5818
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Kidney Stones
Keywords: Ureteral Stent; Kidney Stones
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ureteral stent placement is one of the most common procedures performed within urology. The stents are generally placed for relief of obstruction or to prevent obstruction following a urological procedure. Most patients with ureteral stents will eventually form stent encrustations. However, patients form these encrustations at dramatically different degrees and rates ranging from no encrustation at 1 year of stenting to severe encrustation in just a few weeks. The purpose of this study is to determine if the degree of encrustation on a stent for any given patient can be predicted based on 24 hour urine parameters prior to stent placement, with the stent in place and after stent removal.

Patients who will be receiving stents for other urological reasons will have a 24 hour urine sample collected before stent placement, while the stent is in place and after the stent has been removed. The parameters examined in the 24 hour urine collected will then be compared to the amount of encrustation there is on the stent to see if there is any correlation between the two.

ELIGIBILITY:
Inclusion Criteria:

* Patient at UCI
* Scheduled to undergo surgery (standard of care) where ureteral stent will be placed

Exclusion Criteria:

* minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who will undergo surgery where a ureteral stent will likely be placed will be offered enrollment into this study.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Clayman, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States